CLINICAL TRIAL: NCT05221424
Title: Investigation of The Effect of Training Given According to Roy Adaptation Model On Adaptation to The Disease in Patients With Hypertension
Brief Title: Roy Adaptation Model in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Cihat Demirel, Lecturer, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 206195
Record Dates: First submitted 2022-01-07; First posted 2022-02-03 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-01

CONDITIONS: Hypertension; Patient Engagement; Nurse-Patient Relations
Keywords: Roy adaptation model; patient training; adaptation; hypertension; nursing
MeSH Terms: conditions — Hypertension; Patient Participation | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: This study was conducted as a single-blind randomized controlled study with pretest-posttest
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Experimental): MARS, PAIS-SR and Patient Information Form, containing data about the patient and the disease were applied to each patient in the experimental group during pretest. Then, the individual training was given to each patient by giving the "Hypertension Training Booklet" prepared in line with the Roy Adaptation Model. The training period lasted for averagely 45-50 minutes for each patient. After the training, the patients were called by phone at least once a week, every week for four weeks and reminder information was obtained and their follow-ups were made. One month after the training, post-test data were applied to the patients. In the posttest phase; MARS, PAIS-SR and the questions containing lifestyle changes were repeated and their follow-ups were then terminated.
  Interventions: Other: Patient Education
- No Intervention (No Intervention): • MARS, PAIS-SR and Patient Information Form containing data about the patient and the disease were applied to each patient in the control group in the pretest. Without giving any training to the patients in the control group, only the patients were called at least once a week, every week for four weeks and their health status was examined. One month after the collection of initial data, posttest data were applied to the patients. In the posttest phase; MARS, PAIS-SR and the questions containing lifestyle changes were repeated and then their follow-ups were terminated. After the follow-up, the training prepared in line with Roy Adaptation Model was applied to the voluntary patients and the training booklet was given to them.

INTERVENTIONS:
Other: Patient Education — The training program about hypertension prepared according to the Roy Adaptation Model was performed in a room in the cardiology outpatient clinic of a state hospital. The training content was shaped according to 4 (four) basic areas of the Roy Adaptation Model (physiological field, self-concept field, role function field and interdependence field). The training taught to each patient individually and interactively with the support of powerpoint presentation lasted for averagely 45-50 minutes. A "Hypertension Training Booklet" was prepared according to the Roy Adaptation Model in order to be used during the training and to strengthen the training.
  Arms: Active Comparator

SUMMARY:
The aim of this study was to determine the effect of training given according to the Roy Adaptation Model on medical treatment and physiological, psychological and social adaptation to the disease in individuals with hypertension.

DETAILED DESCRIPTION:
Despite effective and available antihypertensive drugs, the studies showed that less than half of patients with hypertension received antihypertensive therapy and only 1 out of 3 people (less than 20%) had blood pressure control. One of the most important factors in controlling blood pressure in patients with hypertension is the patients' adherence to treatment. Non-adherence to treatment in chronic diseases is considered as a public health problem that increases mortality rates and the economic burden of the disease.

In order to prevent and control hypertension, the importance of non-medical strategies, including lifestyle changes is also emphasized. Lifestyle changes have an important role in increasing treatment and controlling symptoms in hypertensive patients and it is recommended as the first step in managing blood pressure. The most important reason for the failure in the management of hypertension is the patient profile which does not carry out lifestyle changes in parallel with treatment. In this type of patient profile, problems are experienced in the patient's adherence to treatment and it becomes difficult to control blood pressure. Good adaptation to lifestyle changes can reduce the medication needs, lead to a positive effect on cardiovascular risk factors and play an important role for the patient to provide contribution to his/her own treatment.

The non-adherence of hypertensive patients is quite common during their lifestyle changes depending on the disease and during the medication use. Some of the patients stop taking their medications and some do not use their medication regularly. Increasing adherence is the most important factor in success. One of the best ways to increase adherence is to involve the patient in decisions about treatment strategies. One of the factors affecting the adherence to treatment in hypertensive patients is the lack of information about the disease and treatment. For this reason, it is important to increase the awareness and knowledge of patients about the risks associated with blood pressure control in particular. It is possible for hypertensive patients to have knowledge about the disease and treatment, comply with the lifestyle changes and thus control the blood pressure through the training given to the patient. The training and monitoring programs applied for hypertensive patients are one of the best practices that enables the patient to adapt to the disease, control blood pressure and respond to medical treatment faster and live with the disease.

In order for hypertensive patients to comply with the treatment and to implement lifestyle changes, nurses, who are the closest healthcare professionals, have important responsibilities and duties. In the studies, it has been revealed that the interventions applied under the supervision of nurses increase medication adherence. The nursing models, which act as a guide in professional nursing practices and are used in professional development, patient care, and patient training, provide great convenience and assistance in the holistic assessment of the patient. By using models, the problems in the application can be identified by determining the basic concepts of care and the correlation between the concepts and training can be given within this framework by developing solutions for these problems.

In recent years, the use of nursing models in the researches and the patient care management draws a lot of interest in Turkey. One of the models used commonly in the profession is the Roy Adaptation Model (RAM). The purpose of RAM is to provide adaptation for a person to his/her environmental stimuli through adaptive shape methods. According to RAM, individuals should provide and develop their physical and psychological adaptations. This model identifies the reasons of non-adherence to disease and treatment (main and background causes, other stimuli) through an accurate investigation of different individual aspects (for example: physiological aspects, self-perception, role-playing and independence). Thus, it is stated to be helpful in designing a comprehensive training program in order to develop healthy behaviors and comply with the lifestyle changes. Some studies in Turkey showed that the use of RAM increased the adaptation in patients with essential hypertension, increased medication adherence in patients who were followed up with diagnosis of ruptured ectopic pregnancies, and provided positive effects on the diabetes care profile in diabetic individuals. Only one study was found that did not publish when this study was planned, but was seen to be published recently, and evaluating the training given to hypertensive patients using RAM on hypertension management and medical adherence. However, the literature review performed in different databases revealed that there was no study evaluating the effects of training given according to RAM on the disease and psychosocial adjustment in patients with hypertension. For this reason, we assumed that training given by using RAM could cause adherence to medical treatment and disease in the experimental group compared to the control group.

The aim of this study is to evaluate the effects of training given according to Roy Adaptation Model on the disease and psychosocial adjustment in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with hypertension for at least 6 months
* being 18 years old and over
* not having any communication problem
* having no mental confusion or other psychiatric problems
* being literate in Turkish and knowing how to speak Turkish
* being voluntary to participate in the study.

Exclusion Criteria:

* being under 18 years of age
* having cognitive problems
* not wanting to participate in the study
* participating in a similar training program before
* deciding to withdraw the study
* being unable to complete the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-05-27 (Actual)

PRIMARY OUTCOMES:
Medication Adherence Rating Scale (MARS) | 4 weeks after
  In the scale, there are a total of 10 questions that can be answered as yes or no. Negative answers are calculated as 0 point while positive answers are calculated as 1 point. These questions evaluate the patients' adherence to and attitude towards the treatment within the last week. Low score indicates poor adherence to the treatment while high scores indicates high adherence to the treatment.
Psychosocial Adjustment to Illness-Self-Report Scale (PAIS-SR) | 4 weeks after
  The scale contains 46 questions in 7 psychosocial adjustment fields. Psychosocial adjustment fields are "Health Care Orientation" (Part 1), "Vocational Environment" (Part 2), "Domestic Environment" (Part 3), "Sexual Relationships" (Part 4), "Extended Family Relationships" (Part 5), "Social Environment" (Part 6) and "Psychological Distress" (Part 7). The positive statement given to the question is scored with "0" point while negative statement is scored with "3" points. The lowest and highest scores of the scale are 0 and 138 points. In the scale, scores below 35 indicate "good psychosocial adjustment", scores between 35-51 points indicate "moderate psychosocial adjustment", scores above 51 indicate "poor psychosocial adjustment"

CONTACTS AND LOCATIONS:
Locations (1):
- Muş Alparslan University, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: no time limit
Access Criteria: All data
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT05221424/SAP_000.pdf